CLINICAL TRIAL: NCT03279289
Title: Randomised, Multicentre, Phase II Pilot Study to Assess the Efficacy and Safety of Treatment With FOLFIRI-aflibercept Compared to Initial Treatment With FOLFIRI-aflibercept (for 6 Cycles) Followed by Maintenance With 5FU-aflibercept, in an Elderly Population With Metastatic Colorectal Cancer (mCRC) After Failure of an Oxaliplatin-based Regimen
Brief Title: Study to Assess the Efficacy and Safety of Treatment With FOLFIRI-aflibercept Compared to Initial Treatment With FOLFIRI-aflibercept (for 6 Cycles) Followed by Maintenance With 5FU-aflibercept, in an Elderly Population With mCRC After Failure of an Oxaliplatin-based Regimen
Acronym: AFEMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTD-16-03
Record Dates: First submitted 2017-08-03; First posted 2017-09-12 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: FOLFIRI; aflibercept; 5-FU; oxaliplatin; elderly; metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — aflibercept; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): INDUCTION PHASE: 6 cycles of FOLFIRI + aflibercept MAINTENANCE PHASE: 5FU/LV + aflibercept
  Interventions: Drug: Aflibercept; Drug: Irinotecan; Drug: folinic acid (dl racemic); Drug: 5Fluorouracil; Drug: 5-FU
- Group B (Active Comparator): FOLFIRI + aflibercept
  Interventions: Drug: Aflibercept; Drug: Irinotecan; Drug: folinic acid (dl racemic); Drug: 5Fluorouracil; Drug: 5-FU

INTERVENTIONS:
Drug: Aflibercept — 4 mg/kg administered intravenous infusion on day 1
Drug: Irinotecan — 180 mg/m2 intravenous infusion
Drug: folinic acid (dl racemic) — 400 mg/m2 intravenous infusion
Drug: 5Fluorouracil — 400 mg/m2 intravenous bolus
Drug: 5-FU — 2400 mg/m2 continuous intravenous infusion over 46 hours

SUMMARY:
The purpose of this study is to assess the efficacy and safety of treatment with FOLFIRI-aflibercept compared to initial treatment with FOLFIRI-aflibercept (for 6 cycles) followed by maintenance with 5FU-aflibercept, in an elderly population with metastatic colorectal cancer (mCRC) after failure of an oxaliplatin-based regimen

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent, and willing and able to comply with protocol requirements,
2. Histologically proven adenocarcinoma of the colon and/or rectum,
3. Existence of at least one measurable unidimensional lesion using CT or MRI based on the RECIST criteria, version 1.1
4. Patients with metastatic colorectal cancer (mCRC) that is resistant to or has progressed after a first line oxaliplatin-containing regimen for metastatic disease.
5. Age ≥70 years
6. World Health Organization (WHO) Performance status (PS) 0-2,
7. Hematological status: neutrophils (ANC) ≥1.5x109 /L; platelets ≥100x109 /L; haemoglobin ≥9 g/dL
8. Adequate renal function: Creatinine clearance ≥50 mL/min as calculated using the Cockcroft-Gault equation.
9. Adequate liver function: serum bilirubin ≤1.5 x upper normal limit (ULN), alkaline phosphatase (ALP) <5xULN
10. Proteinuria <2+ (dipstick urinalysis) or ≤1g/24hour.
11. Regular follow-up feasible.
12. Male patients with a partner of childbearing potential must agree to use contraception in addition to having their partner use another contraceptive method during the trial.

Exclusion Criteria:

1. Uncontrolled hypercalcemia,
2. Pre-existing permanent neuropathy (NCI grade >2)
3. Uncontrolled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg), or history of hypertensive crisis, or hypertensive encephalopathy,
4. Concomitant protocol unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, immunotherapy),
5. Treatment with any other investigational medicinal product within 28 days prior to study entry.
6. Other serious and uncontrolled non-malignant disease,
7. History or evidence upon physical examination of CNS metastasis unless adequately treated (e.g. non irradiated CNS metastasis, seizure not controlled with standard medical therapy),
8. Patients classified as fragile or delicate according to the following criteria:

   1. Dependence in one or more activities of daily living according to the Katz Index of Independence in Activities of Daily Living (ADL) scale
   2. Three or more comorbidities when assessing the presence of the following processes: congestive heart failure; heart valve disease; coronary artery disease; chronic (obstructive or restrictive) pulmonary disease; cerebrovascular disease; peripheral neuropathy, chronic kidney failure; hypertension; diabetes; concomitant cancers; collagen vascular disease; chronic liver disease; and disabling arthritis
   3. Presence of geriatric syndromes: moderate-severe dementia; delirium in stressful situations (urinary or respiratory tract infection, angina or drugs); moderate-severe depression that interferes with the patient's usual activity; frequent falls (three or more per month); inattentiveness (who could help you in the event of an emergency?); urinary incontinence in the absence of stress, infection, diuretics or prostatic hyperplasia; faecal incontinence in the absence of diarrhoea or laxatives; osteoporotic fractures of large bones or vertebral compression fractures
9. Known Gilbert's syndrome
10. Intolerance to atropine sulfate or loperamide
11. Known dihydropyrimidine dehydrogenase deficiency
12. Treatment with CYP3A4 inducers unless discontinued > 7 days prior to inclusion
13. Any of the following in 3 months prior to inclusion: grade 3-4 gastrointestinal bleeding (unless due to resected tumor), treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, or diverticulitis.
14. Other concomitant or previous malignancy, except: i/ adequately treated insitu carcinoma of the uterine cervix, ii/ basal or squamous cell carcinoma of the skin, iii/ cancer in complete remission for >5 years,
15. Any other serious and uncontrolled non-malignant disease, major surgery or traumatic injury within the last 28 days
16. Patients with known allergy to any excipient to study drugs,
17. History of myocardial infarction and/or stroke within 6 months prior to inclusion, NYHA class III and IV congestive heart failure
18. Bowel obstruction.
19. Less than 28 days elapsed from prior radiotherapy
20. Patients with pernicious anemia or other megaloblastic anemias due to vitamin B12 deficiency
21. Patients with severe infections

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 170 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 48 months

SECONDARY OUTCOMES:
Objective response rate based on the RECIST criteria | 48 months
Disease control rate | 48 months
Depth of response | 48 months
Time to progression | 48 months
Time to treatment failure | 48 months
Overall survival | 48 months
Incidence and severity of AEs CTCAE v4.03 criteria | 48 months
Incidence of dose adjustments and compliance | 48 months
VES-13 score (Vulnerable Elders Survey) as the utility measure for health deterioration | 48 months

OTHER OUTCOMES:
Biomarkers in serum and tumour tissue associated with cell and tumour growth and/or involved in the mechanism of action of FOLFIRI+aflibercept and their correlation with efficacy parameters | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Pilar García Alfonso, Study Chair — Hospital Universitario Gregorio Marañón; Javier Sastre Valera, Study Chair — Hospital Universitario Clínico San Carlos
Locations (1):
- Spanish Cooperative Group for Digestive Tumour Therapy (TTD), Madrid, Spain

IPD SHARING:
Plan to Share IPD: No